CLINICAL TRIAL: NCT02617381
Title: Pre-operative Haemorrhagic Risk Screening, Using a Standardized Questionnaire Before Scheduled Surgeries.
Acronym: HEMORISQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K140901
Record Dates: First submitted 2015-11-19; First posted 2015-12-01 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Pre-operative Haemorrhagic Risk
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- questionnaire (Experimental): assessing the sensitivity and specificity of a simple structured questionnaire
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — assessing the sensitivity and specificity of a simple structured questionnaire

SUMMARY:
"This is not a validation study of a questionnaire. This is a multicenter diagnostic study, assessing the sensitivity and specificity of a simple structured questionnaire, to identify patients requiring further haemostatic investigations, in pre-operative patients. This study will also allow for the assessment of the sensitivity and specificity of the routine care strategy.

All patients are recruited during the pre-anaesthesia visit by an anaesthesiologist, in different anaesthetic sectors each day of the week, so that different types of surgery are represented.

Each day (from Monday to Friday), the first 2 eligible patients will be offered to take part in the study.

Routine care strategy is not modified by the study protocol. In addition, the simple structured questionnaire will be completed by the patient with a research assistant after the pre-operative consultation As recommended in diagnostic studies, the gold standard (see secondary endpoint paragraph) will be performed consistently in all patients to avoid verification bias.

The improvement of screening for the need of further investigations by use of the questionnaire compared to routine care will be measured counting how many patients are adequately reclassified with the questionnaire compared to the routine care strategy, regarding the gold standard (using the Net Reclassification Index)."

DETAILED DESCRIPTION:
"Screening for the need of an extensive haematological investigation in order to determine the existence of inherited or acquired haemostatic abnormalities at the pre-anaesthesia visit is part of a routinely used strategy to prevent perioperative haemorrhagic complications. In France, this screening is mainly based on a basic set of haemostatic tests: prothrombin time (PT), activated partial thromboplastin time (aPTT) and platelet count (PC). When these tests are abnormal, the patient may undergo a more complete set of haemostatic tests and, if needed, be referred to a haematologist for advice. Nevertheless, all published studies have pointed out the scarce efficacy of preoperative PT/aPTT/PC testing for hemorrhagic risk assessment.

Therefore, in 2011 several professional societies have advised AGAINST using this strategy and advocated its replacement by a structured questionnaire for the screening of the need of further haemostatic investigations (to validate or not an increased risk of perioperative haemorrhage). Nevertheless, the performance of a screening strategy relying on such a structured questionnaire has never been studied in the pre-anaesthesia context. This probably explains why many anaesthesiologists still continue to prescribe PT/aPTT/PC to detect haemostatic abnormalities and don't use any questionnaire.

Thus, our hypothesis is that a validated structured and simple questionnaire is an accurate screening strategy to determine patients requiring further haemostatic investigations in the preoperative setting.

One of the main reasons for the non compliance with the guidance advising against the use of screening haemostatic tests (PT/aPTT/PC) for the identification of patients with potential haemorrhagic risk is probably related to the fact that the alternative strategy proposed to anaesthesiologists (the use of a structured questionnaire) has never been investigated before in the context of the pre-anaesthesia visit. Therefore, the present project would estimate the diagnostic performance (sensitivity and specificity) of a simple structured questionnaire to identify patients requiring further haemostatic investigations (i.e. patients for whom further haemostatic investigations would conclude to an increase haemorrhagic risk). The innovative approach of the project is related to: (i) the choice of a simple structured questionnaire, specifically conceived to be used at the pre-anaesthesia visit; (ii) a study design that takes into account the needs of the final users (the anaesthesiologist and the surgical team).

To estimate the diagnostic accuracy of a questionnaire at the pre-anaesthesia visit, to identify patients requiring further haemostatic investigations for haemorrhagic risk assessment as defined by a full haemostatic investigation (i.e. patients for whom full haemostatic investigations would conclude to an increase haemorrhagic risk)

* To estimate the diagnostic accuracy (specificity, sensibility and likelihood ratios) of the current routine care strategy at the pre-anaesthesia visit (i.e. no structured questionnaire, and prescription of further haematological tests at the sole discretion of the anaesthesiologist) to identify patients requiring further haemostatic investigations for HgR as defined by the gold standard (a full haemostatic investigation).
* To measure the improvement in the identification of patients requiring further haemostatic investigations for HgR assessment using a simple structured questionnaire, compared to usual care, in pre-operative patients (i.e. to describe how many patients are adequately reclassified by using the questionnaire).
* To describe how many patients had a major peri-operative bleeding event with respect to the answers to the simple structured questionnaire."

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at the pre-anaesthesia visit by an anaesthesiologist before any scheduled intervention (except for cardiac, vascular, hepatic, obstetrical surgery, since these procedures are associated with a high HgR; neurosurgery is also excluded, due to fatal or functional consequences in case of small volume blood loss).
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Patients under long term antiplatelet and/or anticoagulant therapy
* Not French speaker
* Not affiliated to any social security covering

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Simple structured questionnaire | 3 months
  To estimate the diagnostic accuracy (specificity, sensibility and likelihood ratios) of a simple structured questionnaire at the pre-anaesthesia visit, to identify patients requiring further haemostatic investigations for haemorrhagic risk (HgR) assessment as defined by the gold standard (a full haemostatic investigation), i.e. patients for whom further haemostatic investigations would conclude to an increase haemorrhagic risk.

SECONDARY OUTCOMES:
Use of the Net Reclassification Improvement Index (NRI) | 3 months
  The diagnostic classification provided by the strategy based on the questionnaire compared to that based on hemostasis screening tests will be evaluated by Net Reclassification Improvement Index (NRI)

CONTACTS AND LOCATIONS:
Overall Officials: Dan LONGROIS, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided